CLINICAL TRIAL: NCT06415149
Title: High-Power, Short-Duration Ablation in Treatment of Patients With Atrial Fibrillation
Acronym: HPSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: People's Friendship University of Russia (Other)
Collaborators: City Clinical Hospital No.1 named after N.I. Pirogov (Other)
Responsible Party: Principal Investigator, afsoon fayez, Dr., People's Friendship University of Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27711
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: high-power, short-duration; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power short duration ablation with 50 W (Experimental): Group 1 (n=95): pulmonary vein isolation for treatment of atrial fibrillation was performed with power of 50 watts in Ia subgroup (n=55) AI (ablation index) was 400-450 arbitrary units (au) for the posterior wall and 500-550 au for the anterior wall, in Ib (n=40) AI was 400-450 au for the posterior wall and 450-500 au for the anterior wall.
  Interventions: Procedure: High power short duration ablation with 50 W
- High power short duration ablation with 45 W (Experimental): Group 2 (n=90): Pulmonary vein islolation was performed at a power of 45 watts, in IIa subgroup (n=50) with target AI of 400-450 au for the posterior wall and 500-550 au for the anterior wall in IIb (n=40) AI of 400-450 au for the posterior wall and 450-500 au for the anterior wall.
  Interventions: Procedure: High power short duration ablation with 45 W

INTERVENTIONS:
Procedure: High power short duration ablation with 50 W — Group 1 (n=95): pulmonary vein isolation for treatment of atrial fibrillation was performed with power of 50 watts in Ia subgroup (n=55) AI (ablation index) was 400-450 arbitrary units (au) for the posterior wall and 500-550 au for the anterior wall, in Ib (n=40) AI was 400-450 au for the posterior wall and 450-500 au for the anterior wall.
  Arms: High power short duration ablation with 50 W
Procedure: High power short duration ablation with 45 W — Group 2 (n=90): Pulmonary vein islolation was performed at a power of 45 watts, in IIa subgroup (n=50) with target AI of 400-450 au for the posterior wall and 500-550 au for the anterior wall in IIb (n=40) AI of 400-450 au for the posterior wall and 450-500 au for the anterior wall.
  Arms: High power short duration ablation with 45 W

SUMMARY:
Atrial fibrillation (AF) stands as the most common type of cardiac arrhythmia. The frequency of AF in the overall population is 1-2%, with the incidence rate increasing with age from 0.5% in the 40-50 years old to 5-15% in those aged 80. [According to current recommendations for catheter ablation (CA) in patients with AF, the isolation of the pulmonary veins (PV) is a pivotal aspect of treating this arrhythmia. Despite recent advancements, 20-45% of patients experience recurrences after PV isolation. According to the study by Wasmer K. et al., it was demonstrated that most patients with recurrent AF after PVI showed at least one reconnected vein during redo procedures. The primary cause of recurrences is the restoration of conduction, attributed to endurable isolation (non-transmural, intermittent RF). Numerous approaches have been presented to enhance the outcomes of surgical treatment for AF, such as the CLOSE protocol and Ablation Index (AI) . CLOSE protocol represents an approach aimed at isolating the PV ostia through precise continuous (distance between points ≤ 6 mm) radiofrequency intervention, achieving target ablation index values of ≥ 400au for the posterior wall and ≥ 500au for the anterior wall. The Ablation Index is a marker of quality lesion formation, providing a visual representation of the lesion based on the integration of power, contact force, and time parameters, which is displayed on the CARTO® 3 system (Biosense Webster).

Throughout radiofrequency ablation, electromagnetic energy undergoes conversion into thermal energy, leading to tissue damage and temperature elevation. The temperature elevation process encompasses two stages: resistive heating, impacting surface tissues (1-2mm), and conductive heating, which facilitates the transfer of heat from surface tissues to underlying tissues.

In the presence of good catheter-endocardium contact (25%), only 9% of the power is effectively delivered to the endocardium. For instance, at a power level of 30 watts and optimal contact (25%) with the endocardium, merely 2.7 watts are transferred to the endocardial tissue. When applying 30 watts of power for 30 seconds, a total energy delivery of 900 joules occurs, with only 90 joules being imparted to the endocardium. Similarly, at 50 watts for 10 seconds, only 45 joules of energy are transmitted to the endocardium. When operating at 10 watts, the catheter temperature elevates by 13°C. Consequently, at 30 watts, the temperature reaches 39°C, and at 50 watts, it rises to 65°C. The formation of an irreversible lesion necessitates a temperature exceeding 50°C. During standard radiofrequency ablation (RFA) procedures with power settings ranging from 20 to 45 watts and a duration of 20 to 60 seconds, the formation of ablation points predominantly occurs during the conductive heating phase.

High power short duration ablation (HPSD) is an approach that reduces the conductive heating phase while increasing the resistive heating phase. This results in an expanded area of lesion, facilitating the formation of transmural lesions in the atrial myocardium with irreversible tissue damage and reduced risk to surrounding structures, such as thermal injury to the esophagus.

The strategy of HPSD ablation was developed to overcome limitations of the traditional approach. However, much remains unknown regarding the safety and effectiveness of this approach. Additionally, the question for the optimal interventional treatment method for atrial fibrillation (AF) and the selection of the optimal RF energy for pulmonary vein isolation still require confirmation. This forms the basis for our research objective.

DETAILED DESCRIPTION:
The research was a multi-center retrospective blind randomized controlled trial between 2021 and 2023. A comprehensive sample of 185 participants was enrolled in the study and categorized into 2 cohorts, each of which was further subdivided into two subgroups. Patients were enrolled in the study after providing informed consent. In the first group (n=95), PVI was performed with power of 50 watts in Ia subgroup (n=55) AI was 400-450 arbitrary units (au) for the posterior wall and 500-550 au for the anterior wall, in Ib (n=40) AI was 400-450 au for the posterior wall and 450-500 au for the anterior wall. In the second group (n=90), PVI was performed at a power of 45 watts, in IIa (n=50) with target AI of 400-450 au for the posterior wall and 500-550 au for the anterior wall in IIb (n=40) AI of 400-450 au for the posterior wall and 450-500 au for the anterior wall.

Assessment of conduction block was performed 20 minutes after RFA using a twenty-pole diagnostic electrode (Lasso, Biosense Webster, USA).

ELIGIBILITY:
Inclusion Criteria:

Symptomatic atrial fibrillation (AF) or resistance to at least one antiarrhythmic drug from the first or third group of antiarrhythmic drugs.

Exclusion Criteria:

1. Left atrial thrombosis
2. significant coronary artery disease requiring revascularization
3. valvular heart disease requiring surgical correction
4. acute infectious diseases
5. severe heart failure (NYHA class IV) or left ventricular ejection fraction (LVEF) <35%,
6. history of stroke within the past 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Interoperative outcomes | During ablation
  1-Radiofrequency (RF) ablation duration from start of first pulmonary vein isolation to end of 2-the last lesion.
  3-Total Procedure duration. 4-First pass PVI. 5-Interoperative complications. 6-Total RF energy delivery. 7-Number of RF lesions required for PVI. 8-Freedom from Atrial Fibrillation.
Blinded period | 1- 3 months after ablation
  1. The proportion of patients maintaining Freedom from Atrial Fibrillation.
  2. Overall Complication rate.

SECONDARY OUTCOMES:
Long-term outcomes | 6 -12 months
  1. The proportion of patients maintaining Freedom from Atrial Fibrillation.
  2. The proportion of patients with PV reconnection seen at repeat EP study.

CONTACTS AND LOCATIONS:
Locations (1):
- People's friendship university of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fayez A. , Safonov N. V., Steklov A. S., Faybushevich A. G., Baranovich V. Y. HIGH POWER SHORT DURATION ABLATION USING ABLATION INDEX (AI) IN PATIENTS WITH ATRIAL FIBRILATION // Современная наука: актуальные проблемы теории и практики. Серия: Естественные и Технические Науки. -2023. -№02. -С. 244-250 DOI 10.37882/2223-2966.2023.02.37
- See also: Related Info — http://www.nauteh-journal.ru/index.php/3/2023/%E2%84%9602/6eeb3f6b-3db1-4629-a415-ba018dbd9cbf?lang=en_EN